CLINICAL TRIAL: NCT01425320
Title: Pharmacokinetics Study of Dapsone-Adapalene Fixed Combination Gel in Acne
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was never initiated due to company decision. No study subjects were ever enrolled or dosed.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 225678-003
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone; Gels; Adapalene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fixed Combination dapsone/adapalene Formulation A Gel (Experimental): Study medication will be applied once daily for 14 days to the face, upper chest, upper back, and shoulders.
  Interventions: Drug: Fixed Combination dapsone/adapalene Formulation A Gel
- Fixed Combination dapsone/adapalene Formulation B Gel (Experimental): Study medication will be applied once daily for 14 days to the face, upper chest, upper back, and shoulders.
  Interventions: Drug: Fixed Combination dapsone/adapalene Formulation B Gel
- dapsone 5% gel (ACZONE®) (Active Comparator): Study medication will be applied twice daily for 14 days to the face, upper chest, upper back, and shoulders.
  Interventions: Drug: dapsone 5% gel
- adapalene 0.3% gel (Differin®) (Active Comparator): Study medication will be applied once daily for 14 days to the face, upper chest, upper back, and shoulders.
  Interventions: Drug: adapalene 0.3% gel

INTERVENTIONS:
Drug: Fixed Combination dapsone/adapalene Formulation A Gel — Study medication will be applied once daily for 14 days to the face, upper chest, upper back, and shoulders.
  Arms: Fixed Combination dapsone/adapalene Formulation A Gel
Drug: Fixed Combination dapsone/adapalene Formulation B Gel — Study medication will be applied once daily for 14 days to the face, upper chest, upper back, and shoulders.
  Arms: Fixed Combination dapsone/adapalene Formulation B Gel
Drug: dapsone 5% gel — Study medication will be applied twice daily for 14 days to the face, upper chest, upper back, and shoulders.
  Other Names: ACZONE®
  Arms: dapsone 5% gel (ACZONE®)
Drug: adapalene 0.3% gel — Study medication will be applied once daily for 14 days to the face, upper chest, upper back, and shoulders.
  Other Names: Differin®
  Arms: adapalene 0.3% gel (Differin®)

SUMMARY:
This study will investigate the pharmacokinetics, safety and tolerability of dapsone and adapalene following topical administration of 2 formulations of dapsone/adapalene fixed combination gel, dapsone 5% gel (ACZONE®), and adapalene 0.3% gel (Differin®) in subjects with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Moderate acne on the face
* Willing to avoid swimming during the study
* Willing to avoid excessive sunlight and ultraviolet light (e.g., tanning beds)during the study
* Willing to avoid moisturizers, sunscreens, cosmetics, and chemical peels during the study

Exclusion Criteria:

* Severe cystic acne
* Use of topical or oral retinoids within 4 weeks
* Use of isotretinoin within 3 months
* Use of dapsone or adapalene within 3 months
* Anticipated need to engage in activities/exercise that would cause profuse sweating
* Donated blood or equivalent blood loss within 90 days

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Plasma Levels of Dapsone | Day 1
Plasma Levels of Dapsone | Day 14
Plasma Levels of Adapalene | Day 1
Plasma Levels of Adapalene | Day 14

SECONDARY OUTCOMES:
Local Dermal Tolerability Rating Using a 4-Point Scale | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan